CLINICAL TRIAL: NCT02108574
Title: A Double-blind, Placebo-controlled, Randomized Single-centre Crossover Park Study Assessing Rhinix™ Nasal Filters
Brief Title: Efficacy Park Study Assessing Rhinix™ Nasal Filters for Hay Fever
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Rhinix ApS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1401
Record Dates: First submitted 2014-03-18; First posted 2014-04-09 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Filter (Placebo Comparator): Placebo device
  Interventions: Device: Placebo Filter
- Rhinix Nasal Filter (Active Comparator): Actual Rhinix Nasal Filter
  Interventions: Device: Rhinix Nasal Filter

INTERVENTIONS:
Device: Placebo Filter
  Arms: Placebo Filter
Device: Rhinix Nasal Filter
  Arms: Rhinix Nasal Filter

SUMMARY:
This study will evaluate the effects of RHINIX™ nasal filters on seasonal allergic rhinitis (hay fever) in a park setting.

DETAILED DESCRIPTION:
The study will include 100 participants with grass allergy and will look at the efficacy and usability of RHINIX™ nasal filters on hay fever in a randomized, double-blind, placebo-controlled, crossover design.

ELIGIBILITY:
Inclusion Criteria:

* History of seasonal allergic rhinitis (SAR) for a minimum of 2 years before study entry. Documented by a positive skin test (wheal > 3mm) within 12 months of study enrolment.
* Written informed consent
* Must be able to complete the study
* Reliable anticonception for fertile women
* FEV1 higher than 70 % of predicted value
* Positive grass IgE blood sample higher or equal to 0,7 kU/L

Exclusion Criteria:

* Improper fit of the Rhinix™ device
* Nasal septal deviation
* Retrospective TNSS for last summer < 3
* Positive pregnancy test for fertile women
* Inadequate washout periods in regards to park study appointments (intranasal or systemic corticosteroids (1month), intranasal cromolyn (2 weeks), intranasal or systemic decongestants (3 days), intranasal or systemic antihistamines (3 days), Loratadine (10 days)).
* Rhinitis medicamentosa
* Use of long acting anti-histamines.
* Documented evidence of acute or cronic sinusitis, as determined by the individual investigator.
* FEV1 lower than 70 % of predicted value
* Subjects with nasal conditions likely to affect the outcome of the study in the opinion of the investigator, i.e. anterior nasal septum deviation, nasal septal perforations, nasal polyps, chronic nasal obstruction or other nasal diseases.
* Receipt of immunotherapy with grass pollen within the previous 10 years (at least two rounds of treatment).
* Women who are breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To assess the change in daily Total Nasal Symptom Score (TNSS) between Rhinix™ and placebo | 11.00-17.00 with recordings at 30. minute increments.
  Baseline recording at 09.00 Run-in recordings from 09.30-11.00 Daily Total Nasal Symptom Score evaluated from 11.00-17.00 with the last recording at 17.00, recordings at 30 minute increments.
  Total Nasal Symptom Score is the sum of 4 symptoms (runny nose, blocked nose, itchy nose and sneezing) which are each evaluated on a scale of 0=none, 1=mild, 2=moderate, 3=severe symptoms

SECONDARY OUTCOMES:
To assess the change in Daily Throat Irritation between Rhinix™ and placebo | 11.00-17.00 with hourly increments
  Baseline recording at 09.00 Run-in recording at. 10.00 Daily Throat Irritation evaluated from 11.00-17.00 with the last recording at 17.00, recordings at hourly increments.
  Daily Throat Irritation is the sum of 6 symptom ratings on a Visual Analogue Scale.
To assess the correlation between maximum TNSS and difference in Daily TNSS | 11.00-17.00 at 30 minute increments
  Daily TNSS is described in the Primary Efficacy Endpoint. Maximum TNSS is the single highest TNSS between 11.00 and 17.00
  The correlation will be graphically shown using a Bland-Altman plot.
Change in Daily TNSS for subgroup | 11.00-17.00 at 30 minute increments
  Subgroup analysis of change in daily TNSS between RHINIX and placebo for the subjects with at least one rating of TNSS ≥ 6 on at least one of the two study days.
  See primary outcome measure for more details.

CONTACTS AND LOCATIONS:
Overall Officials: Torben Sigsgaard, Professor, Principal Investigator — Aarhus University, School of Public Health, Dept. of Environmental & Occupational Medicine
Locations (1):
- Aarhus University, School of Public Health, Department of Environmental & Occupational Medicine, Aarhus C, Denmark

REFERENCES:
- [Derived] Kenney P, Hilberg O, Laursen AC, Peel RG, Sigsgaard T. Preventive effect of nasal filters on allergic rhinitis: A randomized, double-blind, placebo-controlled crossover park study. J Allergy Clin Immunol. 2015 Dec;136(6):1566-1572.e5. doi: 10.1016/j.jaci.2015.05.015. Epub 2015 Jun 30. PMID 26141263